CLINICAL TRIAL: NCT04484181
Title: A Randomized Double-blind Trial Evaluating the Live Birth Rate After Transfer of Embryos Cultured in Time Lapse Incubator Compared With Conventional Incubator: Embryoselect
Brief Title: What Embryoselection for What Chance of Success ? EmbryoSelect Study
Acronym: EmbryoSelect
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Programme Hospitalier de Recherche Clinique Inter-Régionale (PHRC-I) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CHUBX 2019/50
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Infertility
Keywords: Embryo; In vitro Fertilization; Selection, Time lapse; Single embryo transfer
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: In the two arms, embryos were cultured and selected for fresh transfer. For the standard incubation group, the selection for transfer was based on morphological criteria. In the TLT group, the selection for transfer was based on morphological and kinetic criteria (with the use of an algorithm).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Embryo culture in time lapse technology (TLT) (Experimental): In the TLT group, the selection for transfer was based on morphological and kinetic criteria (with the use of an algorithm). Embryos will be cultured and selected for fresh transfer.
  Interventions: Other: Embryo culture in time lapse technology (TLT)
- Embryo culture in conventional incubator (Active Comparator): For the standard incubation group, the selection for transfer was based on morphological criteria. Embryos will be cultured and selected for fresh transfer.
  Interventions: Other: Embryo culture in conventional incubator

INTERVENTIONS:
Other: Embryo culture in time lapse technology (TLT) — In the TLT group, the selection for transfer was based on morphological and kinetic criteria (with the use of an algorithm). Embryos will be cultured and selected for fresh transfer.
  Arms: Embryo culture in time lapse technology (TLT)
Other: Embryo culture in conventional incubator — For the standard incubation group, the selection for transfer will be based on morphological criteria. Embryos will be cultured and selected for fresh transfer.
  Arms: Embryo culture in conventional incubator

SUMMARY:
The aim of the research is to evaluate the results of the first in vitro fertilization (IVF) attempt according to the type of embryo culture. From the fertilization to the day 2 transfer, embryos are cultured in standard incubator or in a time lapse technology (TLT). TLT offers an uninterrupted culture environment with a morphokinetic evaluation, whereas culture in standard incubator involves discontinuous morphological embryo evaluation. The principal objective is to compare the live birth rate after the fresh embryo transfer, in a cohort of women less than 39 years-old.

DETAILED DESCRIPTION:
Embryo evaluation and selection is fundamental in clinical IVF in order to obtain a live birth in a shorter delay as possible, but minimizing the risk of multiple pregnancies. TLT was introduced few years ago in clinical practice and allows the continuous follow up of the embryo development. In IVF centers, embryos are preferentially cultured in TL system with undisturbed environmental conditions. This provides information about the development of the embryos in time intervals of 15min and adds kinetic criteria for embryo evaluation and selection. In conventional incubator, the follow up of embryo development consists in 3 static time point observations. Many reviews and observational studies have discussed the value of time-lapse monitoring but it is as yet unclear, however, whether the TLT improves the results of IVF. It has been suggested that the clinical benefits of applying new technologies should be verified and documented by randomized controlled trials. Moreover, the cumulative live birth rate and the delay for conception were rarely reported. The study aims to evaluate the results of the first IVF attempts comparing classical embryo culture in standard incubator and embryo culture and follow up in TLT. The hypothesis is that the undisturbed culture and the selection based on continuous time-lapse images improve the results of the single embryo fresh transfer and increase the cumulative live birth rate. Patients will be randomized the day of the puncture for the type of culture: standard incubation or TLT. The results of the fresh and successive vitrified-warmed embryo transfer will be prospectively collect and patients will be followed until live birth. The attempt will be considered ended after a live birth, if all the frozen embryos are transferred, after 24 months follow up or after surrender.

ELIGIBILITY:
Inclusion Criteria:

* first IVF/ICSI attempt with fresh transfer,
* women ≥18 years-old and <39 years-old,
* signed informed consent

Exclusion Criteria:

* attempts with donor,
* comprehension problem,
* frozen gametes,
* BMI>35 kg/m2,
* history of 3 or more miscarriages,
* uterine pathology,
* serodiscordant patients

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | Month 9
  Live birth rate per punction after the first single embryo fresh transfer. The live birth will be collected 9 months after the first positive pregnancy test

SECONDARY OUTCOMES:
Cumulative live birth rate | Month 9
  Cumulative live birth rate of the attempt (fresh transfer and vitrified-warmed embryo transfers until live birth or use of all vitrified embryos)
Clinical pregnancy rate | Week 6
  Clinical pregnancy rate (cardiac activity at 6 weeks of amenorrhea) per punction and cumulated
Ongoing pregnancy rate | Week 24
  Ongoing pregnancy rate (at more than 24 weeks of amenorrhea) per punction and cumulated
Delay to obtain a live birth | Month 9
  Delay to obtain a live birth (= number of transfers to obtain a live birth)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - clinique Belharra, Bayonne
  - CHU Bordeaux, Bordeaux

IPD SHARING:
Plan to Share IPD: No